CLINICAL TRIAL: NCT02581020
Title: A Follow-up Study to Assess the Durability of Response and Persistence of Resistance to AbbVie's 2 Direct-acting Antiviral Agent (2D) Therapy in Japanese Subjects Who Participated in Phase 2 or 3 Clinical Studies for the Treatment of Chronic Hepatitis C Virus (HCV) Infection
Brief Title: The Durability of Response and Persistence of Resistance to AbbVie's 2 Direct-acting Antiviral Agent (2D) Therapy in Japanese Subjects
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-349
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C; Follow-up; Observation; Japanese
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: Participants who were treated with 2D regimen (ombitasvir/ paritaprevir/ ritonavir) and completed 48 weeks of follow up from the prior Phase 2 or 3 studies conducted in Japan.

SUMMARY:
This study seeks to assess the durability of response and persistence of resistance to ombitasvir/ paritaprevir/ritonavir in Japanese participants who enrolled in a Phase 2 or 3 clinical study with these agents for the treatment of chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Participants treated in Study M12-536 or M13-004 with the 2D regimen (ombitasvir/ paritaprevir/ ritonavir) and completed 48 weeks of follow-up, regardless of SVR achievement.
* Participants who agree to sign the informed consent

Exclusion Criteria:

* Participants treated with a direct-acting antiviral agent (DAA) immediately after Study M12-536 or M13-004.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were treated in Study M12-536 or M13-004 with 2D regimen (ombitasvir/ paritaprevir/ritonavir) and completed 48 weeks of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Hepatitis C virus ribonucleic acid (HCV RNA) levels | 60 months after completion of the 2D treatment in M12-536 or M13-004 study
  HCV RNA levels in plasma

SECONDARY OUTCOMES:
Number of Participants With Resistance-Associated Variants and Phenotypic Resistance to Paritaprevir in Non-structural Viral Protein 3 (NS3) | For approximately 5 years
Number of Participants With Resistance-Associated Variants and Phenotypic Resistance to Ombitasvir in Non-structural Viral Protein 5A (NS5A) | For approximately 5 years
Percentage of participants with hepatocellular carcinoma | Up to 60 month after completion of the 2D treatment in M12-536 or M13-004
Number of participants with serious adverse events (SAEs) | Up to 60 month after completion of the 2D treatment in M132-536 or M13-004 study
  All serious adverse events will be monitored during the observation period.
Hepatitis C virus ribonucleic acid (HCV RNA) levels | 18, 24, 30, 36, 42, 48, 52 months after completion of the 2D treatment in M12-536 or M13-004 study
  HCV RNA levels in plasma

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (53):
- Japan (53):
  - Nagoya City University Hospital /ID# 157439, Nagoya, Aichi-ken
  - Matsuyama Red Cross Hospital /ID# 152125, Matsuyama, Ehime
  - National Hospital Organization Kyushu Medical Center /ID# 161759, Fukuoka, Fukuoka
  - Fukuoka University Hospital /ID# 155965, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 152123, Kurume-shi, Fukuoka
  - Ogaki Municipal Hospital /ID# 158105, Ogaki-shi, Gifu
  - Gunma University Hospital /ID# 158118, Maebashi, Gunma
  - National Hospital Organization Takasaki General Medical Center /ID# 152128, Takasaki-shi, Gunma
  - Hiroshima Red Cross Hospital and Atomic-bomb Survivors Hospital /ID# 152178, Hiroshima, Hiroshima
  - Hiroshima University Hospital /ID# 152232, Hiroshima, Hiroshima
  - Obihiro kosei Hospital /ID# 157437, Obihiro-shi, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 153019, Sapporo, Hokkaido
  - Hitachi General Hospital /ID# 160800, Hitachi-shi, Ibaraki
  - Duplicate_Kanazawa University Hospital /ID# 152226, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital /ID# 153548, Kita-gun, Kagawa-ken
  - Duplicate_Yokohama City University Medical Center /ID# 159474, Yokohama, Kanagawa
  - Yokohama City University Hospital /ID# 165252, Yokohama, Kanagawa
  - Kumamoto Shinto General Hospital /ID# 150061, Kumamoto, Kumamoto
  - Okayama University Hospital /ID# 150060, Okayama, Okayama-ken
  - Osaka City General Hospital /ID# 152126, Osaka, Osaka
  - Japanese Red Cross Osaka Hospital /ID# 155964, Osaka, Osaka
  - Saga University Hospital /ID# 161757, Saga, Saga-ken
  - Saitama Medical University Hospital /ID# 153544, Iruma-gun, Saitama
  - Hamamatsu University Hospital /ID# 152176, Hamamatsu, Shizuoka
  - Dokkyo Medical University Hospital /ID# 152225, Shimotsuga-gun, Tochigi
  - Jichi Medical University Hospital /ID# 153018, Shimotsuke-shi, Tochigi
  - Juntendo University Hospital /ID# 153545, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital /ID# 158121, Bunkyo-ku, Tokyo
  - Toranomon Hospital /ID# 152124, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 152145, Minato-ku, Tokyo
  - Toyama Prefectural Central Hospital /ID# 164156, Toyama, Toyama
  - Yamaguchi University Hospital /ID# 166899, Ube-shi, Yamaguchi
  - University of Yamanashi Hospital /ID# 153547, Chuo-shi, Yamanashi
  - Asakura Medical Association Ho /ID# 155963, Asakura
  - Fukuiken Saiseikai Hospital /ID# 162898, Fukui
  - Gifu Municipal Hospital /ID# 152227, Gifu
  - Gifu Prefectural Genl Med Ctr /ID# 154796, Gifu
  - Ikeda Municipal Hospital /ID# 150062, Ikeda
  - Tokyo Med Uni Ibaraki Med Ctr /ID# 152127, Inashiki
  - Nippon Med Chiba Hokusoh Hosp /ID# 164155, Inzai
  - Kagoshima Uni Med and Dental /ID# 157438, Kagoshima
  - Toranomon Hospital Kajigaya /ID# 152129, Kawasaki
  - Kawasaki Municipal Tama Hospit /ID# 153546, Kawasaki
  - Ehime Prefectural Central Hosp /ID# 158106, Matsuyama
  - Kawasaki Hosp, Kawasaki Med /ID# 152180, Okayama
  - Osaka Hospital /ID# 152177, Osaka
  - Japanese Red Cross Saitama Hos /ID# 166898, Saitama
  - Saiseikai Suita Hospital /ID# 153549, Suita
  - Kagawa Prefectural Central Hos /ID# 152179, Takamatsu
  - Nat Hosp Org Minami Wakayama /ID# 153550, Tanabe
  - Toshiba General Hospital /ID# 152122, Tokyo
  - JP Red Cross Musashino Hosp /ID# 152175, Tokyo
  - Oita University Hospital /ID# 165274, Yufu-shi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — http://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/ombitasvir_P15-349.pdf